CLINICAL TRIAL: NCT06099678
Title: The Effect of Combining Maximal Mental Effort With Elastic Band Training on Strength and Neuromuscular Adaptations in Older Females
Brief Title: Enhancing Strength Gains With the Power of the Mind
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kennesaw State University (Other)
Responsible Party: Principal Investigator, Garrett Hester, Associate Professor of Exercise Science, Kennesaw State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-Harper
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Two intervention groups will perform different types of elastic band training, and a control group will not perform any elastic band training.
Who Masked: Participant
Masking Description: The mental effort aspect of the study will be concealed from subjects, so they will not be aware of any difference between training groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elastic Band Training (Experimental): This group will perform moderate intensity, whole-body elastic band training.
  Interventions: Behavioral: Elastic Band Training
- Elastic Band Training with Maximal Mental Effort (Experimental): This group will perform moderate intensity, whole-body elastic band training with maximal mental effort during muscle contraction.
  Interventions: Behavioral: Elastic Band Training with Maximal Mental Effort
- Control (No Intervention): This group will not perform any training and maintain their regular level of physical activity.

INTERVENTIONS:
Behavioral: Elastic Band Training — This training intervention will be 6 weeks of moderate-intensity elastic band training, including whole-body and isolated muscle exercises.
  Arms: Elastic Band Training
Behavioral: Elastic Band Training with Maximal Mental Effort — This training intervention will be 6 weeks of moderate-intensity elastic band training, including whole-body and isolated muscle exercises, where participants will perform maximal mental effort by imagining maximal muscle contraction during each exercise.
  Arms: Elastic Band Training with Maximal Mental Effort

SUMMARY:
The goal of this clinical trial is to determine the effect of maximal mental effort combined with elastic band training on strength and neuromuscular function in healthy, older females. The main questions it aims to answer are:

* Does elastic band training in combination with maximal mental effort increase strength more than elastic band training alone?
* Does elastic band training in combination with maximal mental effort improve neuromuscular function more than elastic band training alone?

Participants will be randomly assigned to 1 of 3 groups:

* Elastic band training
* Elastic band training with maximal mental effort
* Control

Researchers will compare groups to determine differences in changes in strength, neuromuscular function, and body composition.

DETAILED DESCRIPTION:
Participants in both training groups will perform 6 weeks of moderate intensity, whole-body elastic band training. Participants in the control group will participate in all testing procedures but not perform any training. Participants from both groups will be instructed to maintain their normal physical activity levels and dietary habits.

All training sessions will be home-based and virtually supervised by research personnel. Participants will complete 2 training sessions in the first week and 3 training sessions per week for the remaining 5 weeks. Each training session will last about 45-60 minutes and consist of 7 exercises performed in the same order by each participant, including both multi-joint (chair squat, chest press, leg press, back row) and single-joint (knee extension, knee flexion, elbow flexion) exercises. Participants will perform 12 repetitions for each exercise for the first 3 weeks, then volume will be increased by progressing to 4 sets for the remaining 3 weeks. There will be a 60-second rest interval between sets and a similar tempo will be used between groups.

Both training groups will perform the same training protocol, but participants in the maximal mental effort group will mentally urge their muscles to contract maximally during each repetition. That is, despite using a moderate intensity, participants will imagine the feeling of maximal muscle contraction of the primary muscles during each repetition.

Several measures of strength, neuromuscular function, physical function, and body composition will be measured before and after the training or control period.

ELIGIBILITY:
Inclusion Criteria:

* Between 65-79 years of age
* Female
* Have not engaged in structured exercise for 3 years
* Are not reliant upon a walking aid
* Be able to rise from a chair unassisted
* BMI between 25-33 kg/m²
* Have access to the internet and access to a smartphone or computer with a camera at home

Exclusion Criteria:

* Any history of cardiovascular, cerebrovascular, or metabolic diseases
* Musculoskeletal injury within the past 6 months
* Any condition affecting muscle function
* Uncontrolled hypertension
* Score less than 23 on the Mini-mental State Exam
* Upon starting study, missing more than 2 training session

Ages: 65 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in bicep curl strength as measured by load lifted in pounds | Baseline, Week 7
  Maximum dumbbell load lifted successfully throughout the range of motion of a bicep curl

SECONDARY OUTCOMES:
Change in voluntary activation as measured by ratio of superimposed torque to resting twitch torque | Baseline, Week 7
  Voluntary activation is an estimate of neural drive and is the amplitude of superimposed torque elicited by percutaneous muscle stimulation relative to the resting twitch torque amplitude
Change in handgrip strength as measured in kilograms of force | Baseline, Week 7
  Upper-body strength as measured by a handgrip dynamometer
Change in agonist muscle activation as measured by electromyography amplitude | Baseline, Week 7
  A measure of the capacity at which the muscle is activitated by the nervous system
Change from baseline in isokinetic muscle activation at 6 weeks | Baseline, Week 7
  Electromyography root mean square during isokinetic contraction divided by root mean square during isometric contraction
Change in antagonist co-activation as measured by electromyography amplitude | Baseline, Week 7
  A measure of the capacity at which the antagonist muscle is activated by the nervous system
Change in isometric bicep strength as measured by newton-meters of torque | Baseline, Week 7
  Isometric strength of a muscle
Change in isokinetic bicep strength as measured by newton-meters of torque | Baseline, Week 7
  Dynamic strength of a muscle contracting at a constant velocity
Change in rate of torque development as measured by newton-meters per second | Baseline, Week 7
  A measure of the capacity to increase muscle torque rapidly as determined by the slope of the torque-time curve
Change in walking speed as measured by time taken to walk 6 meters | Baseline, Week 7
  Measure of lower-body physical function
Change in chair rise performance as measured by number of chair rises performed in 30 seconds | Baseline, Week 7
  Measure of lower-body physical function
Change in chair rise power by watts by a linear transducer attached to hip during chair rise test | Baseline, Week 7
  Product of load and velocity as determined on a linear transducer
Change in muscle composition as measured by ultrasound-derived grey-scale analysis | Baseline, Week 7
  Echo-intensity value derived from grey-scale analysis is indicative of amount of non-contractile tissue in muscle
Change in skeletal muscle size as measured by ultrasound-derived cross-sectional | Baseline, Week 7
  Size of a muscle
Change in fat mass as measured by kilograms | Baseline, Week 7
  Amount of fat tissue a person possesses estimated by bioelectrical impedance analysis
Change in fat-free mass as measured by kilograms | Baseline, Week 7
  Amount of non-fat tissue a person possesses estimated by bioelectrical impedance analysis
Change in body fat percentage as measured by fat tissue relative to fat-free tissue | Baseline, Week 7
  Relative amount of body fat a person possesses estimated by bioelectrical impedance analysis
Change in hemoglobin A1c level as measured by blood drop analysis | Baseline, Week 7
  Blood drop analysis, obtained from fingerstick, measure of amount of blood sugar bound to hemoglobin
Change in resting heart rate as measured by beats/min using oscillatory cuff | Baseline, Week 7
  Measure of cardiovascular fitness
Change in resting blood pressure in millimeters of mercury using oscillatory cuff | Baseline, Week 7
  Measure of cardiovascular fitness
Change in general feeling about knee extension and bicep curl exercise | Each exercise session of the 6-week intervention
  From a -5 to +5 on the Affective Feeling Scale
Change in grip width on elastic band as measured by distance of hand placements on band | Baseline, 3 weeks, 5 weeks
  Indication of progression in training intensity

OTHER OUTCOMES:
Change in exercising heart rate | Each exercise session of the 6-week intervention
  A descriptor of the exercise physiological intensity for both training protocols
Change in calorie consumption as measured by kilocalories determined by dietary recall | Baseline, Week 7
  Amount of calories consumed
Change in protein consumption as measured by kilocalories determined by dietary recall | Baseline, Week 7
  Amount of protein consumed
Change in physical activity as measured by daily step count via Garmin Venu SQ smartwatch | Baseline, Week 7
  Measure of physical activity level

CONTACTS AND LOCATIONS:
Overall Officials: Garrett Hester, Ph.D., Principal Investigator — Kennesaw State University
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No